CLINICAL TRIAL: NCT06375980
Title: The Relationship Between Intraoperative Mechanical Power Applied to The Lung and Postoperative Pulmonary Complications in Patients Undergoing Major Abdominal Surgery
Brief Title: Intraoperative Mechanical Power and Ventilation-Associated Lung Injury: Assessing Complications
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arif Timuroğlu, Lead Researcher, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: ANKARA_OR_MP
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Lung Injury; Pulmonary Complication
Keywords: Lung injury; Ventilators, mechanical; Perioperative care; Anesthesia; Risk factors; Ventilator-Induced Lung Injury
MeSH Terms: conditions — Lung Injury; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who developed postoperative pulmonary complications: This cohort consists of patients who developed postoperative pulmonary complications (PPCs). The cohort of patients developing PPCs includes individuals who experienced postoperative hypoxia, atelectasis, bronchospasm, pulmonary infection, pulmonary infiltration, aspiration pneumonia, acute respiratory distress syndrome, pleural effusion, and pulmonary edema. PPCs were assessed using the European Perioperative Clinical Outcome framework.
  Interventions: Other: Intraoperative Mechanical Ventilation Strategies
- patients who did not develop postoperative pulmonary complications .: This cohort comprises patients who did not develop postoperative pulmonary complications (PPCs). The cohort of patients not developing PPCs includes individuals who did not exhibit significant pulmonary complications postoperatively.
  Interventions: Other: Intraoperative Mechanical Ventilation Strategies

INTERVENTIONS:
Other: Intraoperative Mechanical Ventilation Strategies — The intervention involves the management of mechanical ventilation during major abdominal surgery. This includes the adjustment of ventilation parameters such as tidal volume, respiratory rate, peak pressure, positive end-expiratory pressure (PEEP), and inspiratory flow rate. The aim is to optimize ventilation strategies to reduce the risk of postoperative pulmonary complications

SUMMARY:
This study investigates the relationship between intraoperative mechanical power and postoperative pulmonary complications in patients undergoing major abdominal surgery. The investigators record mechanical ventilation parameters and surgical characteristics, assessing the incidence of pulmonary complications within 24 hours postoperatively."

DETAILED DESCRIPTION:
Postoperative pulmonary complications (PPCs) are often underestimated yet remain a leading cause of perioperative morbidity and mortality. These complications encompass postoperative hypoxia, atelectasis, bronchospasm, pulmonary infections, infiltrations, aspiration pneumonia, acute respiratory distress syndrome (ARDS), pleural effusion, and pulmonary edema. They are prevalent and associated with significant costs, prolonging hospital stays, ventilation duration, and ICU admissions, while also increasing mortality and morbidity risks.

Perioperative mechanical ventilation stands as a primary risk factor for the development of postoperative pulmonary complications. Approximately one in four patients with normal lungs will develop some form of lung injury following mechanical ventilation, although much of this damage can be mitigated through the use of appropriate ventilation strategies. A range of pulmonary complications induced by mechanical ventilation is known as ventilator-induced lung injury (VILI).

A growing understanding of the injury mechanism aids researchers in identifying risk factors for lung injury, including tidal volume, respiratory rate, pressures, and flow. Mechanical power, which combines tidal volume, respiratory rate, and airway pressure, has been identified as a potential contributor to VILI. The greater the power, the higher the likelihood of lung injury occurring.

Mechanical power represents the total energy expended over a specific period and is typically expressed in joules per minute (J/min). The equation for mechanical power can help estimate the contribution of different causes of VILI and their variations. This equation can be easily applied in the software of each ventilator. Recent studies have investigated threshold values for mechanical power in relation to ventilator-associated lung injury using the simplified formula found for mechanical power

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients undergoing elective major abdominal surgery
* Patients with ASA (American Society of Anesthesiologists) physical status classification I-IV
* Patients capable of providing voluntary consent

Exclusion Criteria:

* Patients under 18 years of age
* Pregnant individuals
* Those who decline to participate in the study
* Patients requiring reoperation due to surgical complications
* Organ transplant recipients
* Patients who were intubated preoperatively
* Day surgery patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients (aged 18 years and older) scheduled for elective major abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Relationship between mechanical power and postoperative pulmonary complications | Patients were followed for 24 hours postoperatively to evaluate the occurrence of pulmonary complications.
  This study aimed to assess the association between mechanical power and postoperative pulmonary complications. Mechanical power is a crucial parameter for predicting the risk of lung injury related to mechanical ventilation.
  Measurement Tool: Mechanical power calculation based on ventilator parameters. Unit of Measure: Mechanical power expressed in joules per minute (J/min).

CONTACTS AND LOCATIONS:
Overall Officials: Arif Timuroğlu, Study Director — ankara oncology trainig and research hospital
Locations (1):
- Ankara Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel K, Hadian F, Ali A, Broadley G, Evans K, Horder C, Johnstone M, Langlands F, Matthews J, Narayan P, Rallon P, Roberts C, Shah S, Vohra R. Postoperative pulmonary complications following major elective abdominal surgery: a cohort study. Perioper Med (Lond). 2016 May 23;5:10. doi: 10.1186/s13741-016-0037-0. eCollection 2016. PMID 27222707
- [Background] Khan NA, Quan H, Bugar JM, Lemaire JB, Brant R, Ghali WA. Association of postoperative complications with hospital costs and length of stay in a tertiary care center. J Gen Intern Med. 2006 Feb;21(2):177-80. doi: 10.1111/j.1525-1497.2006.00319.x. PMID 16606377
- [Background] Miskovic A, Lumb AB. Postoperative pulmonary complications. Br J Anaesth. 2017 Mar 1;118(3):317-334. doi: 10.1093/bja/aex002. PMID 28186222
- [Background] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Background] Senturk E, Ugur S, Celik Y, Cukurova Z, Asar S, Cakar N. The power of mechanical ventilation may predict mortality in critically ill patients. Minerva Anestesiol. 2023 Jul-Aug;89(7-8):663-670. doi: 10.23736/S0375-9393.23.17080-5. Epub 2023 Apr 20. PMID 37079284